CLINICAL TRIAL: NCT00288873
Title: Characterization of Hyperparathyroidism and Vitamin D Deficiency in Obesity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0509008122
Record Dates: First submitted 2006-02-06; First posted 2006-02-08 (Estimated); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Vitamin D Deficiency; Secondary Hyperparathyroidism; Obesity
Keywords: Vitamin D deficiency; Secondary hyperparathyroidism; Obesity
MeSH Terms: conditions — Vitamin D Deficiency; Hyperparathyroidism, Secondary; Obesity | interventions — Ergocalciferols; Cholecalciferol

INTERVENTIONS:
Drug: Ergocalciferol
Drug: Cholecalciferol

SUMMARY:
Obese persons are known to have elevated levels of parathyroid hormone (PTH) and low levels of vitamin D. These hormones are important in regulation of the body's calcium stores and bone health. We would like to investigate these abnormalities and the accuracy of our current diagnostic tests by comparing results of standard assays for vitamin D and PTH to more specific tests, in obese subjects at baseline and as vitamin D is replaced. We will also compare two standard vitamin D replacement regimens to determine if one is more effective.

This is a pilot study with two parts: Part 1 will compare levels of PTH and vitamin D using two different assays in obese subjects who have normal vitamin D and those who do not. We plan to enroll 20 subjects who have normal vitamin D levels and 40 subjects who have vitamin D insufficiency. All subjects will fill out questionnaires about the amount of calcium and vitamin D in their diet, and their recent sunlight exposure. We will ask for blood samples so that we can measure levels of calcium, vitamin D, albumin, creatinine, glucose, insulin and the different forms of PTH.

Subjects who have vitamin D insufficiency will then be randomized to receive Vitamin D2 or Vitamin D3 in standard doses for eight weeks, in an open label trial. At four and eight weeks, these subjects will fill out the above questionnaires and have the blood tests repeated. For safety purposes, urine calcium will also be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Obese subjects with body mass indices greater than 40 kg/m2 or 35 kg/m2 with other medical conditions secondary to obesity
* Willingness to take vitamin D supplements
* If baseline vitamin D level is >25 ng/ml subjects will be eligible for the control group
* If baseline vitamin D level is <25 ng/ml subjects will be eligible for one of the two vitamin D replacement groups

Exclusion Criteria:

* Hypercalcemia
* Kidney disease
* Liver disease
* Malabsorption
* Prior diagnosis of bone disease
* Medical conditions requiring daily use of calcium, antacids, or medications known to affect bone metabolism or interact with vitamin D
* Hypersensitivity to any formulation of vitamin D

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-02; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Vitamin D (25OHD):RIA and HPLC
Parathyroid hormone (PTH):iPTH and 3rd generation RIA

SECONDARY OUTCOMES:
Parathyroid hormone carboxy terminal fragment levels PTH(7-84)
Ratio of PTH (1-84) to PTH (7-84)
Serum calcium level
Urine calcium level

CONTACTS AND LOCATIONS:
Overall Officials: Emily M Stein, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

REFERENCES:
- [Derived] Stein EM, Strain G, Sinha N, Ortiz D, Pomp A, Dakin G, McMahon DJ, Bockman R, Silverberg SJ. Vitamin D insufficiency prior to bariatric surgery: risk factors and a pilot treatment study. Clin Endocrinol (Oxf). 2009 Aug;71(2):176-83. doi: 10.1111/j.1365-2265.2008.03470.x. Epub 2008 Nov 5. PMID 19018785